CLINICAL TRIAL: NCT02017587
Title: Procurement of Blood Samples for a Biomedical Research Program on T Cell Functional Response to Chronic HBV Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vaccine and Gene Therapy Institute, Florida (Other)
Responsible Party: Sponsor
Other Study IDs: HBV-001
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma/serum PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic HBV: chronic HBV strata: HBV tolerant, Chronic active HBe+ or HBe-, suppressed with antiviral therapy

SUMMARY:
The objective of the study is to procure blood (plasma, serum, RNA and PBMC samples) from approximately 40 chronic HBV for biomedical research program led by VGTI Florida.

DETAILED DESCRIPTION:
During chronic HBV infection, a dynamic balance between viral replication and the host immune response is pivotal to the pathogenesis of liver disease. HBV specific T-cell function is impaired in patients with chronic HBV infection characterized by low levels of antiviral cytokines, impaired cytotoxic T lymphocyte activity, and persistent viremia. However, the mechanism underlying this T-cell malfunction in chronic HBV infection has not been completely understood.

The biomedical research on the samples obtained during this study will include, among other studies, advanced flow cytometry to study the Treg and activation markers, negative regulatory molecules and phenotype of CD4 and CD8 subsets using the extended panel markers developed at VGTI Florida. Additional antibody panels for measuring functional CD4 responses by ICS, DC subsets, activation, and signaling pathways by phos

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic HBV infection documented by presence of HBsAg for at least 12 months currently untreated for HBV infection or under stable antiviral therapy

Exclusion Criteria:

* Prior use of HBV therapeutic vaccine
* Currently treated with interferon alpha or other immune modulator(s)
* Acute HBV infection
* Chronic inactive HBV carrier
* under an acute flare/reactivation of HBV infection defined as symptoms of acute hepatitis and recent elevation of aminotransferase (over 10 x ULN) or bilirubin levels
* Known co-infection with HCV, HDV, and/or HIV
* Under renal dialysis
* For female patients, pregnant or breastfeeding
* Cirrhosis, hepatocellular carcinoma or liver transplantation
* active autoimmune disease including autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
T lymphocyte phenotype and functional response in chronic HBV infection | Baseline
  Phenotype CD4+ and CD8+ subsets - activation markers and negative regulators - CD4+ functional response. Expression of programmed death 1 (PD-1) and its ligand (PD-L1/B7-H1) on viral antigen-specific T-cells

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sterling, MD, Principal Investigator — Virginia Commonwealth University Health System
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States